CLINICAL TRIAL: NCT04915170
Title: Effects of Inspiratory Muscle Training in Adult Patients With Cerebral Palsy
Brief Title: Inspiratory Muscle Training in Cerebral Palsy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, CARLOS MARTIN SANCHEZ, Principal Investigatr, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31052021
Record Dates: First submitted 2021-05-31; First posted 2021-06-07 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Insufficiency
Keywords: aging; cerebral palsy; MANOVA; muscle strength; older adults; physical activity; respiratory exercises
MeSH Terms: conditions — Respiratory Insufficiency; Cerebral Palsy; Motor Activity

STUDY DESIGN:
Intervention Model Description: Patients are assigned randomly to the 2 working groups, each patient only receives one of the two protocols.
Who Masked: Participant, Investigator
Masking Description: The principal investigator doesn´t know the group of the patients until the study ends
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity group (Experimental): Intervention is administrated with an inspiratory muscle trainer (IMT). High intensity group: 10 cycles, 1 minute each one, 40% MIP with IMT. 1 minute to rest between cycles.
  Interventions: Device: Inspiratory muscle training
- Low intensity group (Experimental): Intervention is administrated with an inspiratory muscle trainer (IMT). Low intensity group: 10 cycles, 1 minute each one, 20% MIP with IMT. 1 minute to rest between cycles.
  Interventions: Device: Inspiratory muscle training

INTERVENTIONS:
Device: Inspiratory muscle training — The device incorporate a unidirectional valve independent of flow to guarantee constant resistance and included a specific pressure setting (in cm H2O)

SUMMARY:
To evaluate the effectiveness of two protocols of inspiratory muscle training (IMT) in cerebral palsy patients to improve respiratory strength and spirometric parameters. Low-intensity vs high-intensity resistance training programs. Evaluations: Determination of the maximum inspiratory pressure (MIP) and the maximum expiratory pressure (MEP); spirometry - peak expiratory flow (PEF), forced expiratory volume in first second (FEV1) and clinical evaluations. The participants will be evaluated at the beginning and end of the intervention period. Intervention: There are two groups of patients, one works with low loads (20% MIP) and another with high loads (40% MIP). They train 5 days/week 10 cycles lasting 1 minute. There is a rest of 1 minute between each cycle.

DETAILED DESCRIPTION:
The study was a controlled, randomised, double-blind trial and with allocation concealment. The study protocol was approved by the Bioethics Committee of the University of Salamanca (number of registry 678, 6th October 2021).

Participants:

Institutionalized people with cerebral palsy between 35 and 64 years were included, they were all members of ASPACE Salamanca.

All patients will be asked to carry out the 5-day weekly program, and a recording sheet will be provided to each participant so they will can record the time of each daily respiratory training session. All participants signed an informed consent form.

The patients will be assigned to the two groups randomly. The main researcher doesn´t meet any of the participants until the initial assessment will be carried out.

Intervention:

"High-intensity group". The device incorporates a unidirectional valve independent of flow to guarantee constant resistance and includes a specific pressure setting (in cm H2O).

The intensity of the device will be 40% of MIP. The protocol includes 10 cycles lasting 1 minute. The participants rest for 1 minute between each cycle. In total, the protocol includes 10 minutes of daily respiratory training. The patients will be instructed to inhale with enough force to reach the opening of the valve.

"Low-intensity group".The device incorporates a unidirectional valve independent of flow to guarantee constant resistance and includes a specific pressure setting (in cm H2O).

The intensity of the device will be 20% of MIP. The protocol includes 10 cycles lasting 1 minute. The participants rest for 1 minute between each cycle. In total, the protocol includes 10 minutes of daily respiratory training. The patients will be instructed to inhale with enough force to reach the opening of the valve.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy patients
* Understand the objectives and be able to complete questionaires

Exclusion criteria: the presence of a respiratory disease in the previous month, inability to understand assessment tests or intervention or hemodynamic alterations (heart rate > 150 beats per minute (bpm), systolic blood pressure > 140 millimeters mercury (mmHg) or diastolic blood pressure > 90 mmHg).

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory pressure | 2 minutes
  The evaluation is performed using a pressure transducer, Elka 15, which obtainer each measurement in millibar and converted it into the reference unit of centimeter of water (cm H2O) (1 mbar = 1.01973 cm H2O), following the rules of the American Thoracic Society/European Respiratory Society (ATS / ERS). The procedure was repeated until 3 values were obtained with a difference of less than 5%, and the highest value was used for the analysis.
Maximal expiratory pressure | 2 minutes
  The evaluation is performed using a pressure transducer, Elka 15, which obtainer each measurement in millibar and converted it into the reference unit of centimeter of water (cm H2O) (1 mbar = 1.01973 cm H2O), following the rules of the American Thoracic Society/European Respiratory Society (ATS / ERS). The procedure was repeated until 3 values were obtained with a difference of less than 5%, and the highest value was used for the analysis.

SECONDARY OUTCOMES:
Pulmonary volume | 1 minute
  The evaluation is performed collecting forced expiratory volume in 1 second (FEV1). It was measured using the peak flow device (Asma-1, Vitalograph Ltd, Buckingham, England)
Pulmonary flow | 1 minute
  The evaluation is performed collecting peak expiratory flow (PEF). It was measured using the peak flow device (Asma-1, Vitalograph Ltd, Buckingham, England)

CONTACTS AND LOCATIONS:
Overall Officials: CARLOS MARTIN SANCHEZ, PhD, Principal Investigator — University of Salamanca
Locations (1):
- Carlos Martin Sanchez, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after approving.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After being published.
Access Criteria: Contact the corresponding author.

REFERENCES:
- [Derived] Martin-Sanchez C, Barbero-Iglesias FJ, Amor-Esteban V, Martin-Sanchez M, Martin-Nogueras AM. Inspiratory Muscle Training in Adults With Cerebral Palsy: Long Term Effects: A Double-Blind Randomized, Controlled Trial. Res Nurs Health. 2025 Oct;48(5):545-558. doi: 10.1002/nur.70000. Epub 2025 Jun 20. PMID 40539466